CLINICAL TRIAL: NCT02562248
Title: Improving Anxiety Detection in Pediatrics Using Health Information Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nerissa Bauer, Principal Investigator, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 1508683196; 1508624213 (Other: Indiana University ORA Full Study expedited IRB)
Record Dates: First submitted 2015-09-25; First posted 2015-09-29 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Anxiety; Attention Deficit Hyperactivity Disorder; Disorder, Pediatric
MeSH Terms: conditions — Anxiety Disorders; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): Randomization is at the clinic level. Two clinics will be randomized to receive the revised module to screen for anxiety and ADHD among children who present with parental concern of disruptive behaviors. Parents who have concerns of disruptive behaviors will trigger the module and be administered both the Vanderbilt for ADHD and Screen for Childhood Anxiety Related Emotional Disorders (SCARED) screening tools.
  Interventions: Other: Automated screening for pediatric anxiety
- Control (Active Comparator): Randomization is at the clinic level. Two clinics will be randomized as the control clinics meaning that they will continue to provide care as usual for families who present to the clinic with concerns of disruptive behaviors. Currently, CHICA administers the Vanderbilt for ADHD screening tool.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Automated screening for pediatric anxiety — families receiving care at the intervention clinics with concern for disruptive behaviors will be administered the SCARED tool for anxiety in addition to the Vanderbilt tool for ADHD
  Other Names: SCARED
  Arms: Intervention
Other: Usual Care — families receiving care at the control clinics with concern for disruptive behaviors will be administered the Vanderbilt tool for ADHD only
  Other Names: control
  Arms: Control

SUMMARY:
Inattentive behaviors are a common childhood condition that presents to the general pediatrician. While some of these behaviors are expected during childhood, others need work-up to ensure optimal functioning at home and school. A number of these children ultimately go on to have a mental health conditions, such as ADHD. However, inattentive symptoms represent a broad spectrum of potential behavioral and mental health conditions, such as pediatric anxiety which can masquerade as or co-exist with ADHD. Treatment is quite different and general pediatricians must have ways to facilitate the accurate identification of children needing further work-up and referral. Health information technology can greatly improve pediatricians' ability to identify and refer children with inattentive symptoms for further work-up. This study represents initial work to revise an existing computer decision support system's module for identification of ADHD to include screening questions and prompts for anxiety.

DETAILED DESCRIPTION:
The rapid rate at which childhood mental health and behavioral (MHB) disorders are being identified in primary care practice represents a public health crisis that demands critical examination. Approximately 20% of children and adolescents suffer from a MHB disorder each year. The most commonly recognized childhood MHB disorder is attention deficit hyperactivity disorder (ADHD). Since 2001, when clinical care guidelines were published to help primary care physicians identify ADHD early and initiate psychotropic treatment, ADHD identification has rapidly increased. Children with ADHD are at increased risk of having co-morbid disorders, such as anxiety and depression, oppositional defiant disorder, and learning disabilities, with ADHD symptoms presenting first. Primary care physicians encounter children with symptoms as severe as those in psychiatry clinics; yet a majority in primary care physicians feel ill-equipped to handle MHBs other than ADHD. Two particularly common and vexing problems that can co-occur or masquerade as ADHD are learning disabilities and anxiety. ADHD and anxiety often share behaviors of inattention as the presenting complaint, yet the treatment is quite different. Pediatric anxiety is even more prevalent than ADHD, but often goes undetected and untreated.

In order to improve the detection of ADHD and co-morbidities and prevent undue polypharmacy, validated screening tools are essential in the primary care setting. However, general pediatric practice is fast paced and high volume. Clearly, the ideal diagnostic evaluation of children with symptoms of inattention would involve concurrent administration of validated screening tools for ADHD and anxiety, despite the constraints of a busy pediatric practice. The investigators believe health information technology combined with ongoing quality improvement with input from providers and families can achieve this ideal.

At our institution, we have a computer decision support system, the Child Health Improvement through Computer Automation (CHICA) system that routinely conducts surveillance and screening of commonly encountered pediatric topics. The investigators will build upon the existing ADHD CHICA module, which conducts annual surveillance for inattentive symptoms and integrate validated screening tool for anxiety, associated surveillance items and prompts for the pediatrician to begin to improve the identification of ADHD and anxiety.

Aim 1: Expand and modify the CHICA decision support system to improve the diagnostic processes for screening of children with inattention, including screening in the waiting room, physician prompts, and tailored diagnostic and brief counseling tools.

Aim 2: Improve physician awareness of identification and referral patterns for children presenting with inattentive symptoms by providing run charts for each physician of their screening, referral and medication prescribing patterns paired with facilitated discussion to share strategies to improve diagnostic process and obtain preliminary feedback for future health information technology development of a comprehensive anxiety module.

Aim 3: Examine the effect of the CHICA anxiety module on the diagnostic processes of physicians when screening children with inattentive symptoms.

* Sub-aim 3(a): Evaluate the agreement between positive anxiety screening results obtained by the Vanderbilt and a validated anxiety-specific screening tool.
* Sub-aim 3(b): Evaluate the actions taken by pediatricians when prompted to results of a positive screen.
* Sub-aim 3(c): Compare rates of ICD-9 diagnoses of anxiety and ADHD using billing data and rates of psychotropic medication (stimulants for ADHD versus anxiolytics for anxiety) using e-prescribing data.

ELIGIBILITY:
Inclusion Criteria:

FOR TELEPHONE INTERVIEWS

* Caregivers of children ages 6 to 12 whose parents have concerns of disruptive behavior
* Screening for anxiety is positive using the SCARED tool
* Caregivers must have completed both the SCARED and Vanderbilt tools at the index visit

Exclusion Criteria:

* Primary language is not English or Spanish
* Does not receive medical care at the intervention clinics
* Did not complete both screening tools
* Child did not screen positive for anxiety using the SCARED

FOR PHYSICIAN SATISFACTION

Inclusion criteria:

* all participating providers at all four participating study clinics with CHICA

Exclusion criteria:

* does not provide medical care at any of the four participating study clinics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3267 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Caregiver perception about screening process and satisfaction with index visit | Quarterly, from date of index visit up to 12 weeks
  families will be randomly selected to participate in a one-time telephone interview

SECONDARY OUTCOMES:
Physician satisfaction | annually, from the time module was revised and implemented, up to 2 years
  Physician acceptance of the CHICA anxiety module will be obtained via quantitative surveys addressing physician comfort with anxiety and ADHD identification and acceptance of the anxiety module. These surveys are administered annually as part of ongoing quality improvement. The 30-item survey will include 4 items related specifically to the anxiety module and alterations in the ADHD algorithm. It will require approximately 10 minutes to complete. The survey for will incorporate Likert scales to measure physician comfort with anxiety identification, referral for inattentive behaviors and treatment initiation for anxiety and ADHD. These data will be compared to previously administered surveys that included items capturing physician acceptance of the ADHD module and subsequent management. Results will be aggregated by intervention and control clinics

OTHER OUTCOMES:
Proportion of children screening positive for anxiety | 12 months after implementation of revised module
  Evaluate the agreement between positive anxiety screening results obtained by the Vanderbilt and a validated anxiety-specific screening tool
Actions taken by pediatricians after alert of positive anxiety or ADHD prompt | 12 months after implementation of revised module
  Evaluate the decision making or actions taken by pediatricians when prompted to results of a positive screen. Results will be aggregated by intervention and control clinics
Proportion of ICD-10 Anxiety and ADHD diagnoses | 12 months after implementation of revised module
  Compare rates of ICD-9 diagnoses of anxiety and ADHD using billing data. Results will be aggregated by intervention and control clinics
Comparison of rates of psychotropic medication prescribing for anxiety vs ADHD | 12 months after implementation of revised module
  Rates of psychotropic medication (stimulants for ADHD versus anxiolytics for anxiety) using e-prescribing data. Results will be aggregated by intervention and control clinics

CONTACTS AND LOCATIONS:
Overall Officials: Nerissa S Bauer, MD, MPH, Principal Investigator — Indiana University School of Medicine

IPD SHARING:
Plan to Share IPD: Undecided